CLINICAL TRIAL: NCT01263990
Title: Prospective, Monocentric Pilot Study for the Validation of Stroke Volume by Use of NexFin in Comparison to Different Hemodynamic Monitoring Procedures (Picco2, FloTrac and TEE)
Brief Title: Validation of Stroke Volume Measurement by a New Noninvasive Hemodynamic Monitoring System (NexFin)in Comparison to Different Invasive Procedures as Picco2, FloTrac and TEE
Acronym: VaSNex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Sander, Vice Chair, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VaSNex; EA1/199/10 (Other: Charité Ethics Commission)
Record Dates: First submitted 2010-12-14; First posted 2010-12-21 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Stroke Volume; Mean Arterial Pressure
Keywords: hemodynamic monitoring systems; stroke volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nexfin (No Intervention): Nexfin is used in all patients
  Interventions: Device: NexFin

INTERVENTIONS:
Device: NexFin — noninvasive finger cuff system

SUMMARY:
Main hypothesis: there is no difference between stroke volume measurements recorded by a new noninvasive finger cuff system (NexFin) and invasive hemodynamic monitoring systems as Picco2-system, FloTrac and transesophageal echocardiography

DETAILED DESCRIPTION:
In high risc patients undergoing orthopedic surgery an extended cardiopulmonary observation improves patients safety and postoperative outcome. Therefore invasive procedures as Picco2-system, FloTrac and transesophageal echocardiography (tee) have the advantage to measure or calculate stroke volume. Disadvantage of this treatments is the need for a vascular access with all its complications.

In this study the stroke volume measured by a new noninvasive finger cuff system (NexFin) should be validated in comparison to invasive hemodynamic monitoring systems as Picco2-system, FloTrac and tee.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing orthopedic surgery with need for invasive blood pressure measurements
* age ≥ 18 years
* signed informed consent
* no participation on another interventional study

Exclusion Criteria:

* refusal of participation
* patients who are not able to sign informed consent
* atrial fibrillation with arrhythmia
* peripheral arterial disease > Fontain IIa
* scleroderma
* presence of an arterio-venous shunt on upper limb
* contraindication for femoral arterial vascular access
* contraindication for transesophageal echocardiography
* stage III heart valve defects
* shunt heart defects
* solitary regional anaesthesia
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
stroke volume | preinduction, 3 and 15 minutes after induction, before and after a volume challenge, 30 minutes after induction, end of surgery

SECONDARY OUTCOMES:
mean arterial pressure | preinduction, 3 and 15 minutes after induction, before and after volume challenge, 30 minutes after induction, end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sander, MD, Principal Investigator — Dept. of Anesthesiology Charité Universitaetsmedizin Berlin; Claudia Spies, MD, Study Chair — Dept. of Anesthesiology Charité Universitaetsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum, Berlin, Germany